## INFORMED CONSENT FORM

Online Training to Improve Evidence-based Leadership

Competencies Among Nurse Leaders in Finland: Study

Protocol for a Randomised Feasibility Trial (EVILED-FI)

NCT number: NCT05244512

Approved by The Ethics Committee for Human Sciences at the University of Turku, Health Care Division on 31 May 2022

The ethical number: 12/2022

## SUBJECT'S CONSENT TO PARTICIPATION IN THE STUDY

## Evidence-based leadership in nursing: a randomised feasibility study (EVILEAD-FI)

Psychiatry and Substance Abuse Services of the Department of Social Welfare and Health of the City of Helsinki, Central Finland Hospital District (KSSHP) and University of Turku, Department of Nursing Science

I have been asked to participate in the above-mentioned scientific study, which aims to investigate the effectiveness and preliminary efficacy of the online course on evidence-based nursing leadership. I understand that the course is intended for research participants only.

I have read and understood the research information I have received, and I give my informed consent to participate in the study. I have been adequately informed about the study and the collection, processing and disclosure of data to be carried out in connection with the study. I am aware that the survey data I produce, my login and user data on the Moodle platform, and the learning materials I produce will be used in the study.

I have had the opportunity to receive additional information about the study orally, and I have received adequate answers to all my questions about the study.

I have had sufficient time to consider taking part in the study. I have been adequately informed about the purpose and the conduct of the study, the benefits and risks of the study, and my rights. I have not been pressured or tempted to take part in the study. I am also aware that I have been confirmed by the study coordinator(s) at my hospital and researchers as meeting the inclusion criteria for the study.

I know that my data will be treated confidentially and will not be disclosed to third parties.

I am aware that my personal data may also be processed in the context of an inspection by a domestic or foreign authority, a regular quality control of the research by a person who is not part of the research team (research monitor) and/or a quality assurance activity carried out by a representative of the commissioner.

I understand that participation in this study is voluntary. I understand that I have the right to refuse to participate in the study. I may also discontinue the study or withdraw my consent at any time without giving any reason. I may also withdraw my participation at any stage of the study without giving any reason. I also have the right to withdraw my consent at any time before the end of the study. I am aware that if I discontinue the study or withdraw consent, the data collected about me up to the point of discontinuation and withdrawal of consent will be used as part of the study. I understand that I will not be reimbursed for any expenses incurred for participating in the study.

I confirm my participation in this study, and I voluntarily agree to be a research subject.

[Consent is given electronically in the REDCap system by clicking the option 'I confirm my participation in this study, and I voluntarily agree to be a research subject.']